CLINICAL TRIAL: NCT06327165
Title: Predictability of ANI (Analgesia Nociception Index) for Hypotension After Spinal Anesthesia in Patients Undergoing Cesarean Section
Brief Title: Predictability of ANI (Analgesia Nociception Index) for Spinal Hypotension
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2023-0072
Record Dates: First submitted 2024-03-13; First posted 2024-03-25 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Cesarean Section; Spinal Anesthesia
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pregnant women: Women undergoing cesarean section under spinal anesthesia with ANI monitor applied
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — The ANI monitor calculates heart rate variability mediated by changes in the parasympathetic nervous system.

SUMMARY:
Spinal anesthesia is widely accepted as the anesthetic method of choice for Cesarean section. However, the incidence of spinal hypotension is 50-70%, and the decrease in blood pressure is often rapid and severe. Heart rate variability is influenced by various factors such as the sympathetic nervous system, parasympathetic nervous system, temperature regulation, baroreflex, and endocrine regulation, but high frequency heart rate variability above 0.15 Hz very specifically reflects the parasympathetic nervous system. The ANI monitor calculates heart rate variability mediated by changes in the parasympathetic nervous system. This study aims to determine whether ANI monitor can predict hypotension in patients undergoing a caesarean section under spinal anaesthesia while applying the preemptive vasopressor phenylephrine infusion protocol.

ELIGIBILITY:
Inclusion Criteria:

* full-term parturients undergoing cesarean delivery

Exclusion Criteria:

* emergent surgery, placenta previa, Morbid obesity with a BMI ≥ 40 kg/m2, Gestational age < 36 or ≥ 41 weeks, Contraindications to spinal anesthesia, cardiac arrhythmia, implantable pacemaker, diseases affecting the autoimmune system (such as immune disease or diabetic neuropathy), use of medications affecting ANI monitoring (antimuscarinics, alpha-agonists, beta blockers), illiteracy, or foreigners

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Study Population: ANI monitor will be applied to all patients, but will be covered with black papar so that it could not be observed during anesthesia. ANI data recorded at 1 second intervals will be downloaded at the end of anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
predictive value of ANI monitor for spinal hypotension during cesarean delivery | the occurence of hypotension at (within) 1 hour after spinal anesthesia
  Investigators will determine the predictive power of the ANI score change for the occurrence of hypotension after spinal anesthesia by drawing a receiver operating characteristic (ROC) curve of the change in ANI score (baseline value - minimum value) and calculating the area under the ROC curve.

SECONDARY OUTCOMES:
Optimal cutoff value of ANI level for predicting occurrence of hypotension | the occurence of hypotension at (within) 1 hour after spinal anesthesia
  Investigators will determine the optimal cutoff value of ANI level for predicting hypotension after spinal anesthesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health system, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No